CLINICAL TRIAL: NCT00805012
Title: A Randomized, Multicenter, Phase II Study of Docetaxel and TS-1 Combination as a First-line Treatment in Metastatic or Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Docetaxel and S-1 in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual rate
Sponsor: Seoul National University Hospital (Other)
Collaborators: Clinical Research Center for Solid Tumor, Korea (Other)
Responsible Party: Dae-Seog Heo, Professor, Clinical Research Center for Solid Tumor, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L-0004
Record Dates: First submitted 2008-12-06; First posted 2008-12-09 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: S-1; docetaxel; head and neck cancer; Recurrent or metastatic head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): docetaxel+CDDP
  Interventions: Drug: docetaxel+CDDP
- 2 (Experimental): docetaxel+S-1
  Interventions: Drug: docetaxel+S-1

INTERVENTIONS:
Drug: docetaxel+CDDP — docetaxel+CDDP
  Arms: 1
Drug: docetaxel+S-1 — docetaxel+S-1
  Arms: 2

SUMMARY:
To assess response rate of docetaxel and S-1 combination in metastatic or recurrent head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed HNSCC
* adequate primary site: oral cavity, oropharynx, hypopharynx, nasal cavity, paranasal sinus, other head and neck site (except nasopharynx)
* at least one measurable lesion
* no previous palliative chemotherapy (adjuvant/neoadjuvant chemotherapy and/or radiotherapy longer than 6 months ago is permitted)
* 18 years or older
* ECOG 0 or 1
* adequate laboratory result
* written, informed consent

Exclusion Criteria:

* pregnant or lactating women (negative pregnancy test within 7 days is required for women with potential of child-bearing)
* experimental drug clinical trial within 30 days
* other malignancy (exemption: treated basal cell carcinoma of skin, CIS, cured cancer with disease-free interval with more than 5 years)
* patient with organ transplantation
* grade 2 or more peripheral neuropathy
* grade 2 or more hearing loss
* severe, medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
progression-free survival
duration of response
overall survival
safety

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea